CLINICAL TRIAL: NCT02829411
Title: Testing the Effectiveness of Integrating Relationship Education Into an Existing Workforce Readiness Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MPR-500098-FWCA
Record Dates: First submitted 2016-07-08; First posted 2016-07-12 (Estimated); Last update posted 2021-04-05 (Actual); Status verified 2021-03

CONDITIONS: Marriage; Family Relations

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Employment Services only (Active Comparator): 'Workforce Readiness Program'. job readiness workshop, organized into ten daily sessions over two weeks. The main content of these sessions will be a program-developed workforce readiness training, developed with funding from a DOL Career Pathways Bridge grant.
  Interventions: Behavioral: Workforce Readiness Program
- Employment Services with HMRE content (Experimental): 'Workforce Readiness Program supplemented with Relationship Education': job readiness workshop, organized into ten daily sessions over two weeks. Program will add approximately 17 hours of content from the Within My Reach relationship education curriculum to the two-week job readiness workshop - and add up to eight additional one-hour relationship skills education sessions that customers can attend in the five weeks after completing the initial two-week job readiness workshop
  Interventions: Behavioral: Workforce Readiness Program; Behavioral: Relationship education

INTERVENTIONS:
Behavioral: Workforce Readiness Program — job readiness workshops, organized into ten daily sessions over two weeks.
Behavioral: Relationship education — 25-hours of "Within My Reach" curriculum and relationship skills education sessions
  Arms: Employment Services with HMRE content

SUMMARY:
The project will test the strategy of integrating 25 hours of relationship education into an existing employment program for low-income individuals ages 18-30. It will use a 2-arm randomized controlled trial to test the effect of this full package of services on participants' employment outcomes and relationship outcomes.

DETAILED DESCRIPTION:
The study will examine the programming by FWCA, which currently offers the Career Pathways Bridge program in three locations in St. Louis County in Missouri. The evaluation will test the strategy of integrating relationship education into an existing workforce readiness program. FWCA plans to add approximately 17 hours of content from the Within My Reach relationship education curriculum to the two-week job readiness workshop it offers as part of the Career Pathways Bridge program. Second, FWCA will add up to eight additional one-hour relationship skills education sessions that customers can attend in the five weeks after completing the initial two-week job readiness workshop.

The evaluation will use a 2-arm randomized controlled trial to test the effect of this full package of services on participants' employment outcomes and relationship outcomes. The target population will be low-income individuals ages 18-30 living in St. Louis County, Missouri. The study will aim to enroll 1000 individuals over 2 years. The Metropolitan Employment and Training (MET) Center will be the primary recruitment and service location.

ELIGIBILITY:
Inclusion Criteria:

* disconnected from workforce

Exclusion Criteria:

-

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 909 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2020-12 (Actual)

PRIMARY OUTCOMES:
Perceived romantic relationship skills | 1 year after random assignment
  Six-item scale (α = 0.84) equal to the average level of agreement-from "strongly disagree" (= 1) to "strongly agree" (= 4)-with 6 statements.
Perceived conflict management skills | 1 year after random assignment
  Five-item scale (α = 0.77) equal to the average self-assessment-from "I am bad at this" (= 1) to "I am extremely good at this" (= 4)-of 5 skills.
Support for going slow in romantic relationships | 1 year after random assignment
  Single-item scale equal to the level of agreement-from "strongly disagree" (= 1) to "strongly agree" (= 4)-with the following statement: "People are more likely to succeed in their relationships if they take things slowly."
Disapproval of couple violence | 1 year after random assignment
  Five-item scale (α = 0.77) equal to the average level of disagreement-from "strongly agree" (= 1) to "strongly disagree" (= 4)-with 5 statements.
Any exposure to psychological abuse | 1 year after random assignment
  Binary variable equal to 1 if the respondent indicates that a romantic partner has done any of the following in the past year:
  * Try to keep you from seeing or talking with your friends
  * Make you feel stupid
  * Keep money from you or take your money without asking
  * Made you feel afraid that they might hurt you
Any exposure to physical abuse | 1 year after random assignment
  Binary variable equal to 1 if the respondent indicates that a romantic partner has done any of the following in the past year:
  * Push, shove, or slap you
  * Punch or kick you or beat you up
Any perpetration of physical abuse | 1 year after random assignment
  Binary variable equal to 1 if the respondent indicates that they did any of the following to a romantic partner in the past year:
  * Pushed, shoved, or slapped them
  * Punched, kicked, or beat them up
Involved in an unsteady relationship | 1 year after random assignment
  Binary variable equal to 1 if the respondent reports being involved in an on-again/off-again relationship at the time of the follow-up survey and equal to 0 if the respondent reports being married, engaged, romantically involved on a steady basis, or not in a romantic relationship at the time of the follow-up survey.
Had an unintended pregnancy | 1 year after random assignment
  Binary variable equal to 1 if the respondent reports that they had been/gotten someone pregnant since study enrollment and that they did not want to be/get someone pregnant or the pregnancy came sooner than intended.
Employed or training to improve job prospects | 1 year after random assignment
  Binary variable equal to 1 if the respondent was employed, participating in a job training program, or enrolled in school at the time of the follow-up survey.
Monthly earnings, administrative records | 1 year after random assignment
  Continuous variable constructed from NDNH data that is created by summing quarterly earnings across the four quarters following random assignment and dividing by 12.
Monthly earnings, survey report | 1 year after random assignment
  Continuous variable constructed from survey data that is based on average monthly earnings from all jobs in the first year following study enrollment.
Better off financially now | 1 year after random assignment
  Binary variable equal to 1 if the respondent feels better off financially now than a year ago.
Economic hardship | 1 year after random assignment
  Continuous variable that represents how many of the following six economic hardships the respondent experienced since study enrollment

CONTACTS AND LOCATIONS:
Overall Officials: Brian Goesling, PhD, Principal Investigator — Mathematica Policy Research
Locations (1):
- FWCA, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Undecided